CLINICAL TRIAL: NCT04601545
Title: The Evaluation of the Efficiency of Immersive Virtual Reality Therapy as a Pulmonary Rehabilitation Supporting Method
Brief Title: The Virtual Reality Therapy as a Pulmonary Rehabilitation Supporting Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Foundation for Senior Citizen Activation SIWY DYM (Other)
Responsible Party: Principal Investigator, Joanna Szczepańska-Gieracha, Professor, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VR TierOne PR
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Disease; COPD; Anxiety State; Stress; Depressive Symptoms; Mood Disorders
Keywords: virtual reality; pulmonary rehabilitation; psychotherapy; depression; anxiety; stress; COPD
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Depression; Mood Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR therapy group (Experimental): Pulmonary rehabilitation supplemented by VR therapy
  Interventions: Device: Virtual therapeutic support
- Active Control Group (Active Comparator): Pulmonary rehabilitation supplemented by Schultz Autogenic Training
  Interventions: Behavioral: Pulmonary rehabilitation

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation — Three weeks of pulmonary rehabilitation conducted in an outpatient care facility:
  * 5- time a week for 30 minutes a specific respiratory exercises- relaxation exercises for breathing muscles, exercises to increase breathing, prolonged exhalation exercise, chest percussion
  * 5- time a week for 20-30 min training on a cycle ergometer - until the Heart Rate reaches 60% of the HRmax
  * 5- time a week for 30 minutes a fitness and respiratory exercises - coordination and balance exercises, stretching exercises
  * relaxation by Schultz Autogenic Training. The technique involves the daily practice of sessions that last around 15 minutes. During each session, the practitioner repeats a set of visualisations that induce a state of relaxation.
  Arms: Active Control Group
Device: Virtual therapeutic support — 8 sessions of VR therapy (each of them 20 minutes long). As a virtual reality source, VR Tier One device (Stolgraf®) were used. Thanks to using head mounted display and the phenomenon of total immersion VR therapy provides an intense visual, auditory and kinesthetic stimulation. It can have a calming and mood-improving effect or help the patients recognize their psychological resources and motivate to the rehabilitation process. In the virtual therapeutic garden there are a rich set of symbols and metaphors based on Ericksonian Psychotherapy approach. The most important is the Garden of Revival which symbolizes the patient's health. It used to be full of life and energy, now it is neglected, requires work to be revived. In the therapeutic process day by day, the therapist tells the patient a symbolic story about his/her situation.
  By performing tasks in the virtual garden, the patient becomes an active participant of the therapeutic process and sees the effects his/her work.
  Arms: VR therapy group

SUMMARY:
This study evaluates the effectiveness of virtual reality (VR) therapy in the treatment of depression and anxiety symptoms in patients undergoing the pulmonary rehabilitation. The first study group will receive VR therapy (VR group) as an addition to the traditional pulmonary rehabilitation. The second group (active control group) will receive Schultz Autogenic Training as a standard supplement to the pulmonary treatment. The third group (control group) will undergo only the traditional pulmonary rehabilitation.

DETAILED DESCRIPTION:
Pulmonary rehabilitation leads to the improvement to the physical capacity and overall fitness of the patients with COPD allowing restoration of independence in daily functioning.

Psychological support is required in order to reduce the negative psychological symptoms related to both the pulmonary disease itself and the comorbidities. In this study the investigators want to assess the effectiveness of the virtual reality (VR) therapy compared to standard psychological support (Schultz Autogenic Training).

Thanks to using head mounted display (VR goggles 2018) and the phenomenon of total immersion VR therapy allows to completely separate the patient from the hospital environment, provides an intense visual, auditory and kinesthetic stimulation. Depending on the stage of therapy it can have a calming and mood-improving effect or, in another part of the therapy, it can motivate the patient to the rehabilitation process. The additional aim of the VR therapy is to help the patients regain their emotional balance, let them recognize their psychological resources and trigger the natural recovery mechanisms.

The goals of the project:

1. The evaluation of the influence of VR therapy on the depressive symptoms, the anxiety level and the stress level of the patients undergoing the pulmonary rehabilitation.
2. The comparison of the influence of the VR therapy and Schultz Autogenic Training on the pulmonary rehabilitation process.
3. The evaluation of the pulmonary therapy improvements in patients with and without depressive, anxiety or stress symptoms.

ELIGIBILITY:
Inclusion Criteria:

* COPD;
* Pulmonary rehabilitation conducted in ward settings;
* anxiety symptoms scored 8 and more in HADS-A or depressive symptoms scored 8 and more in HADS-D.

Exclusion Criteria:

* inability to self-complete the research questionnaires;
* presence of the following issues at the time of the examination or in the medical data: disturbances of consciousness, psychotic symptoms or other serious psychiatric disorders;
* initiation of psychiatric treatment during the research project;
* contraindications for virtual therapy (epilepsy, vertigo, eyesight impairment);
* the patient's refusal at any stage of the research project.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 15 minutes
  The Hospital Anxiety and Depression Scale (HADS) is a fourteen-item scale scoring from 0 to 3 for each item. The first seven items relate to anxiety (HADS-A), and the remaining seven items relate to depression (HADS-D). The global scoring ranges from 0 to 42 with a cut-off point of 8/21 for anxiety and 8/21 for depression. The higher the score, the greater anxiety or depression symptoms. HADS will be performed at the beginning and after four weeks of treatment.
Perception of Stress Questionnaire (PSQ) | 30 minutes
  The Perception of Stress Questionnaire (PSQ) is a 27-item scale scoring from 1 to 5 for each item. 21 items examine the level of stress in the area of emotional tension, external stress and intrapsychic stress, and 6 items refer to the lie scale. The global scoring for perception of stress ranges from 21 to 105 with a cut-off point of 60 for high level of perceived stress. The higher the score, the greater the sense of stress. PSQ will be performed at the beginning and after four weeks of treatment.

SECONDARY OUTCOMES:
Six-Minute Walk Test (6MWT) | 10 minutes
  The six-minute walk test measures the distance a patient is able to walk over a total of six minutes on a firm, flat surface. The aim is for the patient to walk as far as possible in six minutes. The patient is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
Spirometry Test | 20 minutes
  The Forced expiratory volume for 1 second (FEV1%pred.) will be analysed as part of the lung function test. The patient is asked to take the deepest breath they can, and then exhale into the sensor as hard as possible, for as long as possible, preferably at least 6 seconds. It is sometimes directly followed by a rapid inhalation, in particular when assessing possible upper airway obstruction. The predicted values will be calculated based on age, weight, and height.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Rutkowski, PhD, Principal Investigator — The Opole University of Technology, Poland; Joanna Szczepańska- Gieracha, Prof, Study Director — University School of Physical Education, Poland; Joanna Szczepańska-Gieracha, Prof, Study Chair — University School of Physical Education, Poland
Locations (2):
- Poland (2):
  - University School of Physical Education, Wroclaw, Lower Silesian Voivodeship
  - Specialist Hospital of the Ministry of Internal Affairs and Administration, Głuchołazy, Opole Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panagioti M, Scott C, Blakemore A, Coventry PA. Overview of the prevalence, impact, and management of depression and anxiety in chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2014 Nov 13;9:1289-306. doi: 10.2147/COPD.S72073. eCollection 2014. PMID 25419126
- [Background] Coventry PA, Bower P, Keyworth C, Kenning C, Knopp J, Garrett C, Hind D, Malpass A, Dickens C. The effect of complex interventions on depression and anxiety in chronic obstructive pulmonary disease: systematic review and meta-analysis. PLoS One. 2013 Apr 5;8(4):e60532. doi: 10.1371/journal.pone.0060532. Print 2013. PMID 23585837
- [Background] Luk EK, Gorelik A, Irving L, Khan F. Effectiveness of cognitive behavioural therapy in a community-based pulmonary rehabilitation programme: A controlled clinical trial. J Rehabil Med. 2017 Mar 6;49(3):264-269. doi: 10.2340/16501977-2189. PMID 28150856
- [Background] da Costa CC, de Azeredo Lermen C, Colombo C, Canterle DB, Machado ML, Kessler A, Teixeira PJ. Effect of a Pulmonary Rehabilitation Program on the levels of anxiety and depression and on the quality of life of patients with chronic obstructive pulmonary disease. Rev Port Pneumol. 2014 Nov-Dec;20(6):299-304. doi: 10.1016/j.rppneu.2014.03.007. Epub 2014 May 27. PMID 24874610
- [Background] Bhandari NJ, Jain T, Marolda C, ZuWallack RL. Comprehensive pulmonary rehabilitation results in clinically meaningful improvements in anxiety and depression in patients with chronic obstructive pulmonary disease. J Cardiopulm Rehabil Prev. 2013 Mar-Apr;33(2):123-7. doi: 10.1097/HCR.0b013e31828254d4. PMID 23399845